CLINICAL TRIAL: NCT05530291
Title: Incidence and Clinical Burden of Erythropoietin Hyporesponsiveness - a Retrospective Database Analysis
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 1517-MA-3435
Record Dates: First submitted 2022-09-05; First posted 2022-09-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; EuCliD; Erythropoietin hyporesponsiveness
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESA hyporesponsive CKD patients: A cohort of patients who meets ESA hyporesponsiveness criteria as well as other common criteria will be created from the Fresenius Medical Care´s proprietary clinical database called EuCliD.
  Interventions: Other: Non-interventional
- ESA responsive CKD patients: A cohort of patients who meets ESA responsiveness criteria as well as other common criteria will be created from the Fresenius Medical Care´s proprietary clinical database called EuCliD.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Epidemiology of anemia associated with chronic kidney disease, rather than to evaluate specific drugs

SUMMARY:
This study consists of two phases. The purpose of phase 1 is to identify incidence and patterns of erythropoiesis-stimulating agent (ESA) hyporesponsiveness and its associated factors in ESA treated patients. The purpose of phase 2 to identify outcomes associated with ESA hyporesponsiveness. Key aspects of the phase 2 study design will entirely depend on the results from phase 1.

DETAILED DESCRIPTION:
This is a retrospective database analysis of patients with anemia associated with chronic kidney disease (CKD) treated with ESAs from January 1st 2015 - December 31st 2021. Data will be derived from European Clinical Database (EuCliD).

ELIGIBILITY:
Inclusion Criteria:

All patients

* Patient has a diagnosis of chronic kidney disease valid between January 1st, 2015, and December 31st, 2021 and is documented in the EuCliD database (incident and prevalent patients)
* Patient who is treated with renal replacement therapy (RRT) (CKD Stage 5) during the study period
* Patient receiving erythropoiesis-stimulating agent (ESA) therapy, within the data collection period having EuCliD data available for a period of the previous 30 days before Index Date but not strictly limited to patients that enter the study period as ESA naïve patients
* Patient having provided consent for secondary use of their data for research purposes
* Patient has a known ESA administration route (intravenous/subcutaneous)
* Patient with a hemoglobin value available at baseline (+/- 20 days allowed) and at least one valid hemoglobin value afterwards
* Patient having at least one body weight value available

Hyporesponsive Cohort

* Patients meeting the hyporesponsive criteria on at least one occasion. The criteria for ESA hyporesponsive will follow the National Institute for Health and Care Excellence, UK (NICE) guidelines:

  * for epoetin alfa, 300 IU/kg/week or more of subcutaneous epoetin or 450 IU/kg/week or more of intravenous epoetin
  * for darbepoetin, dose ≥ 1.5 μg/kg per week

Responsive Cohort

* Patients with all ESA doses lower than those defined by the hyporesponsive criteria

Exclusion Criteria:

* Patient with evidence of hereditary hemolytic anemia (International Classification of Diseases 10th Revision [ICD-10] code D58.9)
* Patient receiving transplant within 6 months prior to Index Date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with anemia of CKD treated with ESA in stage 5D, i.e., on renal replacement therapy (RRT), including extracorporeal RRT and peritoneal dialysis (PD) prevalent as patients in Fresenius Medical Care (FME)'s Nephrocare centers and documented in the EuCliD data base between January 1st 2015 and December 31st 2021.
Sampling Method: Non-Probability Sample
Enrollment: 85259 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Phase 1 Part: Rate of ESA hyporesponsive events | Up to 12 months
  The total number of patients with a new hyporesponsive event in relation to National Institute for Health and Care Excellence, UK (NICE) guidelines within a year after the ESA dose start will be counted as incidence. For deriving the incidence rate, the number of incidence cases will be divided by the sum of the time (days) each patient was observed within this group, totaled for all patients in this ESA subgroup.

SECONDARY OUTCOMES:
Phase 1 Part: Correlation of hyporesponsiveness and patient characteristics over time | Up to 12 months
  Visual representation of hyporesponsiveness and patient characteristics (Hemoglobin [Hb] values, ESA dose, anemia treatment, and NICE defined Hyporesponsiveness) to assess relationship to one another.
Phase 1 Part: Time from the start of ESA dose to the first hyporesponsive event | Up to 12 months
  The time until the first hyporesponsiveness event will be estimated.
Phase 1 Part: Distribution of ESA hyporesponsiveness patients | Up to 12 months
  Hyporesponsive events will be categorized into isolated, intermittent and chronic, and distribution will be evaluated.
Phase 1 Part: Baseline characteristics | Day 1 (start of ESA treatment)
  Demographics and clinical characteristics of patients who developed ESA hyporesponse and those that did not (responders) will be compared.
Phase 1 Part: Characteristics on date of first incidence satisfying hyporesponsiveness criteria | Up to 12 months
  Demographics and clinical characteristics of patients who developed ESA hyporesponse will be compared with a matched control group.
Phase 1 Part: Percentage of ESA hyporesponsiveness in relation to the KDIGO definition | At 12 months
  Percentages in relation to the Kidney Disease: Improving Global Outcomes (KDIGO) definition will be provided for the ESA hypo-responders and the ESA responders.
Phase 1 Part: Percentage of ESA hyporesponsiveness per Clinical Practicability Algorithm | At 12 months
  Percentages per Clinical Practicability Algorithm will be provided for the ESA hyporesponders and the ESA responders.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site DE49001, Bad Homburg, Germany

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Atzinger C, Arens HJ, Neri L, Arkossy O, Garbelli M, Jiletcovici A, Snijder R, Leyland K, Khalife N, Ali M, Feuersenger A. Hyporesponsiveness to Erythropoiesis-Stimulating Agents in Dialysis-Dependent Patients with Anaemia of Chronic Kidney Disease: A Retrospective Observational Study. Adv Ther. 2025 Jan;42(1):471-489. doi: 10.1007/s12325-024-03015-4. Epub 2024 Nov 25. PMID 39581908
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/1517-MA-3435/